CLINICAL TRIAL: NCT06493110
Title: Comparison of Gastric Volumes With Ultrasound in Diabetic and Non-diabetic Term Pregnant Women Before Elective Cesarean Section
Brief Title: Gastric Ultrasound in Term Pregnants
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Feyza Calisir, Assistant professor, Kahramanmaras Sutcu Imam University
Other Study IDs: 2022/26-12
Record Dates: First submitted 2024-03-22; First posted 2024-07-09 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy; Diabetes
Keywords: Gastric ultrasound; Term pregnant; Preoperative fasting
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic term pregnant: 1. Patients with good mental status
  2. Pregnant patients aged ≥18 years
  3. Patients in ASA II-III group
  4. Patients complying with preoperative fasting instructions (at least 6 hours for solids, at least 2 hours for clear liquids)
  5. Term pregnant women (gestational age ≥ 36 weeks)
  6. 50-120kg weight
  7. 150cm height or taller
  8. Have written informed consent
  Interventions: Procedure: Gastric ultrasound
- non-diabetic term pregnant: 1. Patients with good mental status
  2. Pregnant patients aged ≥18 years
  3. Patients in ASA II-III group
  4. Patients complying with preoperative fasting instructions (at least 6 hours for solids, at least 2 hours for clear liquids)
  5. Term pregnant women (gestational age ≥ 36 weeks)
  6. 50-120kg weight
  7. 150cm height or taller
  8. Have written informed consent
  Interventions: Procedure: Gastric ultrasound

INTERVENTIONS:
Procedure: Gastric ultrasound — To compare gastric volumes in standard fasting state before surgery in diabetic and non-diabetic pregnant women by evaluating the gastric antrum with ultrasound.

SUMMARY:
In this study, the investigators aimed to evaluate the gastric antrum with ultrasound and compare gastric volumes in diabetic and non-diabetic pregnant women in the standard fasting state before surgery. The primary aim was qualitative assessment, while secondary objectives included quantitative assessment, comparing gastric volume, aspiration risk, and the effect of preoperative anxiety on stomach contents.

DETAILED DESCRIPTION:
Food residues in the stomach of patients scheduled for surgery are a major risk factor for pulmonary aspiration, leading to significant morbidity and mortality. This risk is particularly critical in pregnant women who may require surgery without proper fasting. National guidelines recommend fasting for 6 hours for solid foods, 4 hours for breast milk, and 2 hours for clear liquids. These guidelines apply equally to adults and children. Pregnant patients scheduled for elective surgery follow the same fasting rules as non-pregnant patients.

Gastroparesis, defined as delayed gastric emptying without mechanical obstruction, affects 30-50% of diabetic (DM) patients. Ultrasound measurement of the gastric antral area can help identify whether the stomach is full in symptomatic patients. Gastric ultrasound is a valuable tool for assessing aspiration risk in pregnant women, especially during emergency surgeries, and has shown promise in fasting non-pregnant patients scheduled for elective surgery.

In this study, the investigators aimed to evaluate the gastric antrum using ultrasound and compare gastric volumes in diabetic and non-diabetic pregnant women in a standard fasting state before surgery. The primary goal was qualitative assessment, with secondary objectives including quantitative assessment, comparing gastric volume, aspiration risk, and the effect of preoperative anxiety on stomach contents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with good mental status
2. Pregnant patients aged ≥18 years
3. Patients in ASA II-III group
4. Patients complying with preoperative fasting instructions (at least 6 hours for solids, at least 2 hours for clear liquids)
5. Term pregnant women (gestational age ≥ 36 weeks)
6. 50-120kg weight
7. 150cm height or taller
8. Written informed consent

Exclusion Criteria:

1. Taking any medication known to accelerate or delay gastric emptying, including (but not limited to) opioid-containing medications and antacids.
2. Gastroesophageal reflux, abnormal anatomy of the upper gastrointestinal tract, previous surgical procedures for the esophagus or upper abdomen, etc. any stomach complaints
3. Pregnant women with term labor or obstetric emergency
4. Twin pregnancy -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This cohort comprised 30 diabetic and 30 non-diabetic individuals. The included participants were mentally healthy, aged 18 and above, classified as ASA II-III according to the American Society of Anesthesiologists, and had a gestational age of 36 weeks or more.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Gastric Antrum Quality | 12 months
  Qualitative evaluation of the gastric antrum using ultrasound: For the qualitative evaluation of the gastric antrum, we used a grading scale where the gastric antrum is classified as Grade 0, 1, or 2. The grading criteria are as follows:
  Grade 0: The stomach appears empty in both supine and right lateral decubitus positions.
  Grade 1: The stomach appears empty in the supine position but shows clear fluid in the right lateral decubitus position.
  Grade 2: Clear fluid is seen in the stomach in both supine and right lateral decubitus positions.

SECONDARY OUTCOMES:
Gastric Volume | 12 months
  Quantitative measurement of gastric volume in milliliters.
Aspiration Risk | 12 months
  Number of participants with a high aspiration risk based on gastric volume.
Preoperative Anxiety Effect | 12 moths
  Measurement of stomach content volume related to preoperative anxiety levels.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KahramanmarasSIU, Kahramanmaraş
  - Kahramanmaraş Sutcu Imam University, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No